CLINICAL TRIAL: NCT07225868
Title: Prepare the Mind: Can Coaching in Goal-directed Behaviour Increase the Success of Cognitive Rehabilitation in People With MS?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Leiden (Other)
Collaborators: Reha Rheinfelden (Other); University at Buffalo (Other)
Responsible Party: Principal Investigator, Marit Ruitenberg, PhD, Universiteit Leiden
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL86331.058.24; OZ2023-017 (Other Grant/Funding Number: Dutch National MS Funds)
Record Dates: First submitted 2025-11-03; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Conscientiousness; Cognitive Rehabilitation; Brain Imaging; Quality of Life
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conscientiousness Coaching (Experimental)
  Interventions: Behavioral: Conscientiousness Coaching Before Cognitive Rehabilitation
- Sham Intervention (Sham Comparator)
  Interventions: Behavioral: Sham Intervention Before Cognitive Rehabilitation

INTERVENTIONS:
Behavioral: Conscientiousness Coaching Before Cognitive Rehabilitation — In this arm, participants complete the conscientiousness coaching before the cognitive rehabilitation. All participants (both arms) will receive 6 weeks of cognitive rehabilitation using BrainHQ (2 times per week, 1 hour each).
  Arms: Conscientiousness Coaching
Behavioral: Sham Intervention Before Cognitive Rehabilitation — In this arm, participants complete the sham intervention before the cognitive rehabilitation. All participants (both arms) will receive 6 weeks of cognitive rehabilitation using BrainHQ (2 times per week, 1 hour each).
  Arms: Sham Intervention

SUMMARY:
People with Multiple Sclerosis (MS) often experience cognitive difficulties such as memory problems, concentration issues, and reduced processing speed. These symptoms can have a negative impact on daily functioning and overall quality of life. Previous research on cognitive rehabilitation has shown that regular training focused on memory and concentration can have positive effects on cognitive functioning, including processing speed, memory, and executive functions that support daily activities. Moreover, fMRI studies (brain scans that measure brain activity) have revealed changes in brain activation following cognitive rehabilitation.

Recently, the idea has emerged that a more personalized approach could improve treatment outcomes. Specifically, researchers have identified a link between personality traits and cognitive functioning. Since every individual is different, current cognitive rehabilitation programs often fail to take these personal differences into account.

In this project, the investigators aim to enhance the effectiveness of cognitive rehabilitation by focusing more closely on individual characteristics through an app-based training program. Participants will complete a 12-week app training prior to a 6-week cognitive rehabilitation program. The first app focuses on mindset training, supported by a coach. Afterwards, all participants will use a second app designed to train processing speed and memory. In addition to cognitive functioning, the investigators will also examine psychological, (neuro)biological, and social changes using questionnaires and fMRI. This research may provide valuable insights into how cognitive functioning and quality of life in people with MS can be improved.

This study is funded by the National MS Fund and is a collaboration between several institutions: the Department of Health, Medical and Neuropsychology at Leiden University (The Netherlands), the University at Buffalo (USA), and Reha Rheinfelden (Switzerland).

DETAILED DESCRIPTION:
Rationale: Cognitive impairment displays a common and impacting symptom in people with multiple sclerosis (PwMS). It has been shown that PwMS benefit from cognitive rehabilitation (CR), but group-effects are mild-to-moderate and effect sizes vary between patients, highlighting the need for including individual factors in investigating CR. It has been shown that PwMS with high conscientiousness, a personality trait that is associated with being well-organised, schema driven, achievement-striving and goal-directed show higher improvement on cognitive functions. Very recent data shows that it is possible to enhance conscientiousness in PwMS and that this increase led to more goal-directed behaviour, decreased depressive symptoms and improvements in QoL.

Objective: To investigate if conscientiousness coaching (C-Coach) before CR will enhance the treatment effects of CR, in which treatment effect is operationalised as improvement from a full comprehensive perspective of well-being of PwMS Study design: This experimental multicentre study in the Netherlands, United States and Switzerland follows a longitudinal, parallel group, controlled design with three assessment sessions including behavioural testing for both study groups and brain imaging in a subsample. Additionally, both groups will undergo either 12-weeks of C-Coach or sham training before six weeks of CR.

Study population: The study population consists of 126 PwMS aged between 18 and 65 years, of which group 1 (N= 63) will undergo C-Coach before CR and group 2 (N= 63) will undergo a sham intervention before CR.

Intervention: All interventions will be performed on mobile devices and can thus be done at home. Group 1 will undergo 12 weeks of C-Coach, which consists of a pre-session and two booster sessions with a coach to explain goals, values and the training application as well as the self-use of the smartphone application C-Coach between sessions to track goals and values. Group 2 will undergo 12 weeks of sham intervention, consisting of a pre-session and two booster sessions with a coach to discuss early life memories and the self-use of the smartphone application Daily Notes to journal about early life memories. Both groups will undergo CR after C-Coach or sham intervention, where they are asked to perform two 60-minutes training sessions per week for the duration of 6 weeks using the CR training application BrainHQ.

Main study parameters/endpoints: Main endpoint will be subjective and objective cognitive changes between baseline and post-intervention on processing speed task and improved cognitive functioning in daily life in PwMS in the intervention group compared to PwMS in the control group. As secondary endpoints, changes between baseline and post-intervention on goal attainment, meaning of life, fatigue, depression, anxiety, cognitive functioning, functional brain networks and social support in PwMS in the intervention group (C-Coach prior to CR) compared to PwMS in the control group (sham intervention prior to CR) will be studied.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The risk of proposed interventions and procedures including MRI scan is negligible, as both can be seen as safe and non-invasive. All participants in the subsample undergoing MRI scans will undergo a detailed screening for MRI contradictions to exclude any risks. The confined space inside the MRI device for the duration of 25 minutes of the scan as well as the time investment of the participant for travel to study location and participation involves some burden for the participants. This study will offer valuable insights in the development of effective cognitive rehabilitation strategies, which will in turn positively impact patients' QoL and their ability to participate in society as they see fit.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed relapsing remitting or secondary progressive MS diagnosis according to the McDonald 2017 criteria
* Expanded Disability Status Scale (EDSS) score < 7
* Relapse free period ≥ 3 months
* Unchanged disease modifying therapy for ≥ 2 months at time of inclusion
* Age 18-65 years
* Language Dutch, English or German for each centre respectively

Exclusion Criteria:

* High conscientiousness, measured with a T score 65 or higher on the BFI-2 subscale for conscientiousness
* Current or prior brain trauma or neurological condition (other than MS)
* Psychiatric disorder that heavily impacts cognitive and/or daily functioning
* Medication intake and/or substance abuse that has an influence on cognitive functioning
* For Dutch subsample undergoing MRI: Contradiction for MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective cognitive changes between baseline and post-intervention | Between baseline and week 18.
  Objective cognitive changes between baseline and post intervention will be assessed using the Symbol Digit Modalities Test assessing information processing speed.
Subjective cognitive changes between baseline and post-intervention | Between baseline and week 18.
  Subjective cognitive changes between baseline and post intervention will be assessed using the Multiple Sclerosis Instrumental Activities of Daily Living Questionnaire.

SECONDARY OUTCOMES:
Changes between baseline and week 18 on meaning of life in the intervention compared to the sham intervention group. | Between baseline and week 18.
  Changes on the Meaning of Life Questionnaire comparing the intervention (C-Coach prior to CR) group with the sham intervention group.
Changes between baseline and week 18 on fatigue in the intervention compared to the sham intervention group. | Between baseline and week 18.
  Changes on the Checklist of Individual Strength comparing the intervention (C-Coach prior to CR) group with the sham intervention group.
Changes between baseline and week 18 on quality of life in the intervention compared to the sham intervention group. | Between baseline and week 18.
  Changes on the 36-Item Short Form Survey comparing the intervention (C-Coach prior to CR) group with the sham intervention group.
Changes between baseline and week 18 on psychological outcomes in the intervention compared to the sham intervention group. | Between baseline and week 18.
  Changes on the Hospital Anxiety and Depression Scale comparing the intervention (C-Coach prior to CR) group with the sham intervention group.
Changes between week 12 and week 18 on goal attainment in the intervention compared to the sham intervention group. | Between week 12 and week 18.
  Changes on the Goal Attainment Scale comparing the intervention (C-Coach prior to CR) group with the sham intervention group.
Changes between baseline and week 18 on multiple sclerosis specific cognitive functioning in the intervention compared to the sham intervention group. | Between baseline and week 18.
  Changes on the Brief International Cognitive Assessment for Multiple Sclerosis comparing the intervention (C-Coach prior to CR) group with the sham intervention group.
Changes between baseline and week 18 on cognitive flexibility in the intervention compared to the sham intervention group. | Between baseline and week 18.
  Changes on the Trail Making Test A and B comparing the intervention (C-Coach prior to CR) group with the sham intervention group.
Changes between baseline and week 18 on verbal fluency in the intervention compared to the sham intervention group. | Between baseline and week 18.
  Changes on the Controlled Oral Word Association Test comparing the intervention (C-Coach prior to CR) group with the sham intervention group.
Changes between baseline and week 18 executive functions in the intervention compared to the sham intervention group. | Between baseline and week 18.
  Changes on the Stroop Test comparing the intervention (C-Coach prior to CR) group with the sham intervention group.
Changes between baseline and week 18 on functional networks in the intervention compared to the sham intervention group. | Between baseline and week 18.
  Changes on functional networks measured with resting state functional magnetic resonance imaging comparing the intervention (C-Coach prior to CR) group with the sham intervention group.
Changes between baseline and week 18 on structural networks in the intervention compared to the sham intervention group. | Between baseline and week 18.
  Changes on Structural networks measured with Diffusion Tensor Imaging comparing the intervention (C-Coach prior to CR) group with the sham intervention group.
Changes between baseline and week 18 on social outcomes in the intervention compared to the sham intervention group. | Between baseline and week 18.
  Changes on the Medical Outcomes Study Social Support Survey comparing the intervention (C-Coach prior to CR) group with the sham intervention group.

OTHER OUTCOMES:
Effect of personality | Between baseline and week 18.
  The effect of baseline trait conscientiousness, neuroticism and personality measured with the Big Five Inventory 2 on all outcomes.
Effect of demographics | Between baseline and week 18.
  The effect of baseline demographic variables, namely age, sex, nationality, and education will be studied on the described outcomes.
Effect of C-Coach | Between baseline and week 12.
  The main and secondary outcomes will be measured at week 12 after C-Coach or sham intervention and before the start of CR in order to replicate previous preliminary findings.
Feedback on C-Coach or sham intervention | At week 18.
  Participants' responses to a Feedback Questionnaire will be examined at week 18, which includes specific questions about the effectiveness and the experience of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke E Hulst, Prof, Principal Investigator — Leiden University; Priska Zuber, PhD, Principal Investigator — Reha Rheinfelden; Ralph HB Benedict, Prof, Principal Investigator — Jacobs School of Medicine and Biomedical Sciences, Neurology, University at Buffalo; Marit FL Ruitenberg, PhD, Principal Investigator — Leiden University
Locations (3):
- Jacobs School of Medicine and Biomedical Sciences, Neurology, University at Buffalo, Buffalo, New York, United States
- Health, Medical and Neuropsychology, Institute of Psychology, Faculty of Behvavioural and Social Siences, Leiden University, Leiden, Netherlands
- Research Department, Reha Rheinfelden, Rheinfelden, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about study and recruitment — https://mindslab.nl/onderzoek/prepare-the-mind/